CLINICAL TRIAL: NCT01573065
Title: Addressing HIV Risk in Young Unhealthy Alcohol Drinkers in the Emergency Department With Rapid HIV Testing and Brief Intervention
Brief Title: HIV Testing and Brief Alcohol Intervention for Young Drinkers in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Lynn E. Fiellin, Associate Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0906005270
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Alcohol Consumption; Sexual Risk Behaviors
Keywords: alcohol consumption; sexual risk behaviors; young, unhealthy drinkers
MeSH Terms: conditions — Alcohol Drinking | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Behavioral: Counseling intervention with rapid HIV testing

INTERVENTIONS:
Behavioral: Counseling intervention with rapid HIV testing — Counseling intervention (modeled after Brief Negotiation Interview and Project RESPECT-2) coupled with rapid HIV testing. Telephone booster at 2 weeks.

SUMMARY:
The purpose of this study was to determine whether a brief counseling intervention coupled with rapid HIV testing was feasible and effective at decreasing alcohol consumption and sexual risk behaviors among young, unhealthy drinkers presenting to the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old;
* engaged in at least one sexual risk behavior in past 90 days;
* alcohol consumption greater than NIAAA guidelines for at-risk drinking;
* unknown or negative HIV status and willing to be tested;
* able to provide contact information for follow-up;
* able to provide written informed consent.

Exclusion Criteria:

* known HIV positive status;
* medically or psychiatrically unstable.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Feasibility | baseline and 2 month follow-up
  number of patients enrolled and retained at 2 months.

SECONDARY OUTCOMES:
Alcohol consumption | baseline vs. 2 month follow-up
  As assessed by the Time Line Follow Back, change in alcohol consumption.
Sexual risk behaviors | baseline vs. 2 month follow-up
  As assessed by an adapted HIV Risk Behaviors Scale, change in sexual risk behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Fiellin, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Emergency Deparmtment, New Haven, Connecticut, United States